CLINICAL TRIAL: NCT02938546
Title: 18F-FDG Metabolism Imaging Monitoring Non-small Cell Lung Cancer Curative Effect of Chemotherapy Multicenter Clinical Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Wenhui XIE, chief physician, Shanghai Chest Hospital
Allocation: Non-Randomized | Model: Factorial | Masking: Double | Purpose: Diagnostic
Other Study IDs: WXIE
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Non-small-cell Lung Cancer
Keywords: Non-small-cell lung cancer; 18F-FDG PET/CT; treatment response assessment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- before therapy (Active Comparator): 18F-FDG PET/CT performed before therapy
  Interventions: Radiation: 18F-FDG
- 3 days after cisplatin chemotherapy and targeted therapy (Experimental): 18F-FDG PET/CT performed 3 days after chemotherapy and targeted therapy
  Interventions: Radiation: 18F-FDG
- longer time after cisplatin chemotherapy and targeted therapy (Experimental): 18F-FDG PET/CT performed before the third cycle chemotherapy and the 7th week targeted therapy
  Interventions: Radiation: 18F-FDG

INTERVENTIONS:
Radiation: 18F-FDG — 18FDG-PET scan was performed 4 weeks before the first administration of therapy or before the third cycle chemotherapy or before the 7th week of targeted therapy and after 3 days chemotherapy and targeted therapy. The lesions were analyzed by nuclear medicine physician and calculate the metabolism response. The size of percent changes was evaluated using the EORTC (European Organization for Research and Treatment of Cancer) PET criteria by oncologist who determine whether the scheme works and the scheme should continue or change. The seleted patients were double blinded to analyse the relationship between metabolism response and chemotherapy response.

SUMMARY:
The subject is going to use 18F-FDG PET/CT to assess different genetic NSCLC metabolism after cisplatin chemotherapy and targeted therapy, define the assessment criteria for the role of 18F-FDG PET/CT in NSCLC treatment respone and at last build multi-centre clinical trial platform of molecular classification and molecular imaging for cancer chemotherapy assessment.

DETAILED DESCRIPTION:
Non-small-cell lung cancer (NSCLC) is the first leading cause of cancer death in the world. Systemic chemotherapy has contributed to the only choice for more than 50% NSCLC patients. The genetic abnormalities lead to different therapy response to the same chemotherapy scheme in NSCLC patients. At present, early assessment and prediction is the key for optimize NSCLC therapy. 18F-FDG PET/CT is a noninvasive cell metabolism reaction molecular imaging technology which can assess cancer glucose metabolism sensitively and react cancer proliferation to some degree. Hence 18F-FDG PET/CT may be used to assess NSCLC therapy response noninvasively. It is a reliable method to individualize NSCLC treatment clinically by define the appropriate metabolism response cut-off values and assess time points of 18F-FDG PET/CT in predicting different genetic NSCLC patients.The subject is going to use 18F-FDG PET/CT to assess different genetic NSCLC metabolism after cisplatin chemotherapy and targeted therapy, define the assessment criteria for the role of 18F-FDG PET/CT in NSCLC treatment respone and at last build multi-centre clinical trial platform of molecular classification and molecular imaging for cancer chemotherapy assessment.

ELIGIBILITY:
Inclusion Criteria:

* pathological biopsy for NSCLC; stage III-IV; plan to palliative chemotherapy (such as neoadjuvant chemotherapy, convention and targeted therapy) due to unable to surgery; not radiation therapy or chemotherapy for 6 months before enrollment; the predictive survival time more than half year;

Exclusion Criteria:

* with diabetes and chest radiotherapy chronic disease; brain metastases patients; with secondary primary maligmant cancer in 5 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-11; Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Glucose metabolism discrepancy of different genotype NSCLC as Assessed by EORTC | 6 years

SECONDARY OUTCOMES:
Different genotype NSCLC metabolic response after treatment as Assessed by EORTC | 6 years

OTHER OUTCOMES:
Time points of predictive specific genotype NSCLC glucose metabolic response by statistics | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Wenhui Xie, PHD, Study Director — Shanghai Chest Hospital of Shanghai Jiao Tong University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zhao Y, Wang H, Shi Y, Cai S, Wu T, Yan G, Cheng S, Cui K, Xi Y, Qi X, Zhang J, Ma W. Comparative effectiveness of combined therapy inhibiting EGFR and VEGF pathways in patients with advanced non-small-cell lung cancer: a meta-analysis of 16 phase II/III randomized trials. Oncotarget. 2017 Jan 24;8(4):7014-7024. doi: 10.18632/oncotarget.12294. PMID 27690345
- [Result] Zhang T, Xie J, Arai S, Wang L, Shi X, Shi N, Ma F, Chen S, Huang L, Yang L, Ma W, Zhang B, Han W, Xia J, Chen H, Zhang Y. The efficacy and safety of anti-PD-1/PD-L1 antibodies for treatment of advanced or refractory cancers: a meta-analysis. Oncotarget. 2016 Nov 8;7(45):73068-73079. doi: 10.18632/oncotarget.12230. PMID 27683031
- [Result] Watanabe K, Shinkai M, Tei Y, Kaneko T. Chemotherapy in Non-Small Cell Lung Cancer Patients Receiving Oxygen Therapy. Oncol Res Treat. 2016;39(10):587-590. doi: 10.1159/000449328. Epub 2016 Sep 15. PMID 27710970
- [Result] Shang J, Ling X, Zhang L, Tang Y, Xiao Z, Cheng Y, Guo B, Gong J, Huang L, Xu H. Comparison of RECIST, EORTC criteria and PERCIST for evaluation of early response to chemotherapy in patients with non-small-cell lung cancer. Eur J Nucl Med Mol Imaging. 2016 Oct;43(11):1945-53. doi: 10.1007/s00259-016-3420-7. Epub 2016 May 28. PMID 27236466
- [Result] Ho TY, Chou PC, Yang CT, Tsang NM, Yen TC. Total lesion glycolysis determined per RECIST 1.1 criteria predicts survival in EGFR mutation-negative patients with advanced lung adenocarcinoma. Clin Nucl Med. 2015 Jun;40(6):e295-9. doi: 10.1097/RLU.0000000000000774. PMID 25783515
- [Result] Lee DH, Kim SK, Lee HY, Lee SY, Park SH, Kim HY, Kang KW, Han JY, Kim HT, Lee JS. Early prediction of response to first-line therapy using integrated 18F-FDG PET/CT for patients with advanced/metastatic non-small cell lung cancer. J Thorac Oncol. 2009 Jul;4(7):816-21. doi: 10.1097/JTO.0b013e3181a99fde. PMID 19487962
- [Result] Huang W, Zhou T, Ma L, Sun H, Gong H, Wang J, Yu J, Li B. Standard uptake value and metabolic tumor volume of (1)(8)F-FDG PET/CT predict short-term outcome early in the course of chemoradiotherapy in advanced non-small cell lung cancer. Eur J Nucl Med Mol Imaging. 2011 Sep;38(9):1628-35. doi: 10.1007/s00259-011-1838-5. Epub 2011 May 27. PMID 21617977
- [Result] Wijesinghe P, Bollig-Fischer A. Lung Cancer Genomics in the Era of Accelerated Targeted Drug Development. Adv Exp Med Biol. 2016;890:1-23. doi: 10.1007/978-3-319-24932-2_1. PMID 26703796
- [Result] Tafe LJ, Pierce KJ, Peterson JD, de Abreu F, Memoli VA, Black CC, Pettus JR, Marotti JD, Gutmann EJ, Liu X, Shirai K, Dragnev KH, Amos CI, Tsongalis GJ. Clinical Genotyping of Non-Small Cell Lung Cancers Using Targeted Next-Generation Sequencing: Utility of Identifying Rare and Co-mutations in Oncogenic Driver Genes. Neoplasia. 2016 Sep;18(9):577-83. doi: 10.1016/j.neo.2016.07.010. PMID 27659017
- [Result] Yuneva MO, Fan TW, Allen TD, Higashi RM, Ferraris DV, Tsukamoto T, Mates JM, Alonso FJ, Wang C, Seo Y, Chen X, Bishop JM. The metabolic profile of tumors depends on both the responsible genetic lesion and tissue type. Cell Metab. 2012 Feb 8;15(2):157-70. doi: 10.1016/j.cmet.2011.12.015. PMID 22326218
- [Result] Masri S, Papagiannakopoulos T, Kinouchi K, Liu Y, Cervantes M, Baldi P, Jacks T, Sassone-Corsi P. Lung Adenocarcinoma Distally Rewires Hepatic Circadian Homeostasis. Cell. 2016 May 5;165(4):896-909. doi: 10.1016/j.cell.2016.04.039. PMID 27153497
- [Result] Dejust S, Morland D, Fabre G, Prevost A, Papathanassiou D. 18F-FDG PET/CT Evaluation of Ceritinib Therapy in Metastatic ALK-Positive Non-small Cell Lung Cancer. Clin Nucl Med. 2016 Nov;41(11):879-880. doi: 10.1097/RLU.0000000000001361. PMID 27607176
- [Result] Manegold C, Dingemans AC, Gray JE, Nakagawa K, Nicolson M, Peters S, Reck M, Wu YL, Brustugun OT, Crino L, Felip E, Fennell D, Garrido P, Huber RM, Marabelle A, Moniuszko M, Mornex F, Novello S, Papotti M, Perol M, Smit EF, Syrigos K, van Meerbeeck JP, van Zandwijk N, Yang JC, Zhou C, Vokes E. The Potential of Combined Immunotherapy and Antiangiogenesis for the Synergistic Treatment of Advanced NSCLC. J Thorac Oncol. 2017 Feb;12(2):194-207. doi: 10.1016/j.jtho.2016.10.003. Epub 2016 Oct 8. PMID 27729297